CLINICAL TRIAL: NCT06058260
Title: Assessment of Cognitive Function and Quality of Life in Thalassemic Children at Sohag University Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mena Gerges Shawky, Resident-pediatric department-sohag hospital university, Sohag University
Other Study IDs: Soh-Med-23-09-07MS
Record Dates: First submitted 2023-09-13; First posted 2023-09-28 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Thalassemia
MeSH Terms: conditions — Thalassemia | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children With Thalassemia (Cases): Hematological Disease which are a heterogeneous group of single gene disorders, inherited in an autosomal recessive manner ( Thalassemia Syndrome )
  Interventions: Other: Pediatric Quality of Life Inventory (questionnaire) and The Stanford-Binet Intelligence Scale fifth edition
- Healthy Children ( Controls ): Healthy Children free from any chronic illness
  Interventions: Other: Pediatric Quality of Life Inventory (questionnaire) and The Stanford-Binet Intelligence Scale fifth edition

INTERVENTIONS:
Other: Pediatric Quality of Life Inventory (questionnaire) and The Stanford-Binet Intelligence Scale fifth edition — Quality of Life Assessment By Pediatric Quality of life Inventory. Cognitive Function Assessment By The Stanford-Binet Intelligence Scale fifth edition.

SUMMARY:
Thalassemia syndromes are a heterogeneous group of single gene disorders, inherited in an autosomal recessive manner ,prevalent among all ethnic groups and in almost every country around the world .

Once a child has been diagnosed as thalassemia, he has to take lifelong treatment , where cure is not attainable and treatment may be prolonged . It is a life-threatening and life-limiting condition that affects the patient clinically and psychologically, so Health-related Quality of Life (HRQOL) is likely to be an essential outcome for these patients.

Quality of life in thalassemic children such as : Repeated visits to hospitals for regular blood transfusion, cost of chelation therapy, repeated laboratory tests for monitoring therapy and for early detection of any complications. also life-long costly therapy along with poor quality of life will have adverse impact on the family.

A better understanding of the factors associated with HRQOL among children with thalassemia could have a direct effect on the development of more suitable clinical, counselling and social support programs to enhance treatment outcomes.

Cognitive dysfunction was Reported either due to the disease or its treatment ,frequent school absences, frequent hospitalizations, and physical and social restrictions lead to cognitive dysfunction . This neurological involvement in thalassemic children is primarily silent, with subclinical manifestations that can only be detected by cognitive assessment tests.

DETAILED DESCRIPTION:
Thalassemia syndromes are a heterogeneous group of single gene disorders, inherited in an autosomal recessive manner ,prevalent among all ethnic groups and in almost every country around the world .

Thalassemias are genetic diseases characterized by a deficit in the production of hemoglobin, the protein contained in red blood cells that transports oxygen in the bloodstream. The disease is qualified as α-thalassemia or β-thalassemia depending on whether the anomaly results from a defect in the synthesis of the alpha (α) chains or beta (β) chains making up the protein.

It is the most prevalent chronic hemolytic anemia in Egypt (85.1%), the carrier rate of thalassemia in 1000 normal subjects was found to be 9-10.2% .

Once a child has been diagnosed as thalassemia, he has to take lifelong treatment , where cure is not attainable and treatment may be prolonged . It is a life-threatening and life-limiting condition that affects the patient clinically and psychologically, so Health-related Quality of Life (HRQOL) is likely to be an essential outcome for these patients.

The principles of treatment have been well defined which include (a) maintaining hemoglobin between 9 and 10 g/dl by repeated packed cell transfusion (b) regular chelation therapy to maintain serum ferritin around 1000 ng/dl (c) preventing the development of complications of the disease or secondary to therapy (d) ensuring normal growth and development . This conventional treatment is required for life-long. The main objective of thalassemia life-long treatment is to maintain good quality of life as close to near normal life. there are many Factor that can affect Quality of life in thalassemic children such as : Repeated visits to hospitals for regular blood transfusion, cost of chelation therapy, repeated laboratory tests for monitoring therapy and for early detection of any complications. also life-long costly therapy along with poor quality of life will have adverse impact on the family.

The assessment of HRQOL in children is essential for the provision of proper care, since it helps in identifying the impact of the disease and treatment on children . A better understanding of the factors associated with HRQOL among children with thalassemia could have a direct effect on the development of more suitable clinical, counselling and social support programs to enhance treatment outcomes.

Cognitive dysfunction was Reported either due to the disease or its treatment ,frequent school absences, frequent hospitalizations, and physical and social restrictions lead to cognitive dysfunction . This neurological involvement in thalassemic children is primarily silent, with subclinical manifestations that can only be detected by cognitive assessment tests.

Previous studies showed significantly different results between patients and controls regarding the intelligence quotient (IQ).

ELIGIBILITY:
Inclusion Criteria:

* All the diagnosed thalassemic children age between 4 and 18 years.

Exclusion Criteria:

* Any other hematological disease.
* Age less than 4 years and more than 18 years.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All the diagnosed thalassemic children age between 4 and 18 years.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-10-20 (Estimated); Primary Completion 2024-10-20 (Estimated); Study Completion 2024-10-20 (Estimated)

PRIMARY OUTCOMES:
The Stanford-Binet Intelligence Scale fifth edition | 12 months
  Assessment of Cognitive Function Minimum Value is 40 Maximum value is 160 Higher scores mean a better outcome
Pediatric Quality of Life Inventory | 12 months
  Assessment of Quality of Life Minimum value is 0 Maximum value is 100 Higher scores mean a better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Choudhry VP. Thalassemia Minor and Major: Current Management. Indian J Pediatr. 2017 Aug;84(8):607-611. doi: 10.1007/s12098-017-2325-1. Epub 2017 Apr 24. PMID 28435994